CLINICAL TRIAL: NCT02550691
Title: Identification of a Biomarker Associated With Cis-duplication of the SMN1 Gene Aiming at Improving the Genetic Counseling in Spinal Muscular Atrophy Families
Brief Title: Identification of a Biomarker Associated With Cis-duplication of the SMN1 Gene
Acronym: BADGES
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Financial sponsor difficulties
Sponsor: University Hospital, Rouen (Other)
Collaborators: Society GENOMIC VISION (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015/092/HP
Record Dates: First submitted 2015-09-14; First posted 2015-09-15 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Spinal Muscular Atrophy
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Subject carrying 3 copies of the SMN1 gene (Experimental): Using blood sampling, use of molecular combing to identify a genomic morse code (GMC) composed of a combination of probes specific of a structural motif on the cis-duplication chromosome.
  Interventions: Procedure: blood sampling
- Subject carrying 2 copies of the SMN1 gene (Other): Using blood sampling, use of molecular combing to identify a genomic morse code (GMC) composed of a combination of probes specific of a structural motif on the cis-duplication chromosome.
  Interventions: Procedure: blood sampling
- Subject carrying 3 copies of the SMN2 gene (Other): Using blood sampling, use of molecular combing to identify a genomic morse code (GMC) composed of a combination of probes specific of a structural motif on the cis-duplication chromosome.
  Interventions: Procedure: blood sampling

INTERVENTIONS:
Procedure: blood sampling — A blood sample will be taken on subject carrying specific genotype

SUMMARY:
Spinal Muscular Atrophy (SMA) is a neuromuscular disorder characterized by loss of motor neurons in the anterior horn of the spinal cord and leading to muscle atrophy. SMA has an autosomal recessive inheritance and affects 1 in 6000 infants with a carrier frequency of 1 in 40. In most cases, it is caused by homozygous gene deletion or gene conversion of the SMN1 gene (0+0 genotype) on 5q11-q13. This genomic region has been duplicated and inverted during evolution. Thus the SMN1 gene has a very homologous copy, called SMN2. Genetic counseling aim at detecting carriers with only one copy of the SMN1 gene (0+1 genotype). SMA carrier testing relies on total copy number quantification of the SMN1 copies by quantitative PCR methods. Nevertheless, cis-duplication of the SMN1 gene on one allele and deletion on the second allele (2+0 genotype) can lead to a misinterpretation as molecular methods show 2 copies of the SMN1 gene and cannot detect the carrier status.

The aim of the study is the characterization of a biomarker specific of the cis-duplication of the SMN1 gene in order to allow the detection of this 2+0 genotype which constitutes a trap for genetic counseling. We will use molecular combing to identify a genomic morse code (GMC) composed of a combination of probes specific of a structural motif on the cis-duplication chromosome. The characterization of this GMC is based on the comparison of two sample groups:

* The test group, with a maximum of 137 individuals carrying 3 copies of the SMN1 gene (suggesting a cis-duplication on one allele)
* The control-1 group, with a maximum of 137 individuals carrying 2 copies of the SMN1 gene

A pilot study performed on 24 samples in the two groups is needed to define the exact sample number necessary for statistical analysis of the study. When the GMC will be characterized, its specificity will be evaluated by testing two sample groups:

* The test group, with 37 individuals carrying 3 copies of the SMN1 gene
* The control-2 group, with 37 individuals carrying 3 copies of the SMN2 gene Molecular combing needs long DNA fibers and usual methods for DNA extraction are not appropriate. This project requires new blood samples for specific DNA extraction.

If this project is successful, during a second project, this GMC will be converted into a simple and cheap PCR-based method. We will then evaluate the sensitivity of this method on our sample collection, notably on individuals with the 2+0 genotype defined by familial genotyping.

ELIGIBILITY:
Inclusion Criteria:

* Adult individual
* Individual with either 2 copies of the SMN1 gene (control-1 group), 3 copies of the SMN1 gene (test group), or 3 copies of the SMN2 gene (control-2 group).
* Individual with a social insurance
* Signed consent form

Exclusion Criteria:

* Pregnant women, nursing women
* Individual without freedom by administrative decision or judicial decision or individual under administrative supervision or legal guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-12-15 (Actual); Primary Completion 2016-07-04 (Actual); Study Completion 2016-07-04 (Actual)

PRIMARY OUTCOMES:
Identification of a genetic signature indicating the presence of one allele with 2 copies in cis of the SMN1 gene. | Day 1

SECONDARY OUTCOMES:
Specificity of a genetic signature | Day 1
  Specificity of a genetic signature will be done using analysis of individual carrying either 3 copies of the SMN1 gene or 3 copies of the SMN2 gene

CONTACTS AND LOCATIONS:
Overall Officials: Thierry FREBOURG, MD, Principal Investigator — University Hospital, Rouen
Locations (2):
- France (2):
  - Nantes University Hospital, Nantes
  - Rouen University Hospital, Rouen